CLINICAL TRIAL: NCT01924247
Title: Prospective Randomized Study to Validate the Effects of an Outpatient Secondary Prevention Program for Stroke Victims With Minor or no Residual Deficits
Brief Title: Study to Validate the Effects of an Outpatient Secondary Prevention Program for Stroke Victims
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Schweizerische Herzstiftung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 090/13
Record Dates: First submitted 2013-08-09; First posted 2013-08-16 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Cerebrovascular Disorders; Stroke; Prevention
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional Arm (Other): Interventional Arm
  Interventions: Behavioral: Outpatient secondary prevention program
- Control Arm (Other): Control Arm: Standard treatment by family physician
  Interventions: Behavioral: Standard treatment by family physician

INTERVENTIONS:
Behavioral: Outpatient secondary prevention program — The comprehensive outpatient program is designed to last for 12 weeks. Participants are treated in groups of 8 or less. Every week there are two days with therapeutic and educational sessions, once with two hours of physical exercise therapy and once with 45 minutes of aerobic ergometer training and one hour of lecture and counseling. On the day with the two hours of physical therapy one of the sessions includes aerobic ergometer training or Nordic walking, and the other session focuses on improvements of fine motor skills, coordination, balance, mobilization, stretching, weight training or breathing. The lectures include three lectures on etiology, diagnosis, treatment and prevention of stroke by a neurologist, one on vascular risk factors by a cardiologist, five on nutrition counseling by nutritionists, two on active and passive smoking cessation and one lecture on psychological coping strategies given by a neuropsychologist.
  Arms: Interventional Arm
Behavioral: Standard treatment by family physician — Standard treatment by family physician.
  Arms: Control Arm

SUMMARY:
Background:

Stroke represents one of the major health problems worldwide, particularly in transitional and industrialized countries. Stroke has a remarkable socioeconomic impact, especially in the ageing population, and therefore stroke prevention is important. Secondary preventive measures and rehabilitation are essential for reduction of recurrent events. However, to date appropriate secondary preventive programs for patients surviving a stroke with minor or no residual deficits have been poorly studied.

Specific aims/projects:

The aim of this study is to validate the effects of an outpatient secondary prevention program on vascular risk factors, adherence to vascular-protective medication, exercise capacity and health related quality of life.

Working Hypothesis:

The outpatient rehabilitation program results in a significant short (3 months) and long-term (1 year) improvement of vascular risk factors, neurological functions, exercise capacity, adherence to vasoprotective medication and health related quality of life.

Experimental design/Methods:

This is a prospective, randomized clinical trial. At least 100 patients will be randomized either to the interventional group or to a group which is treated only by the family physician. All patients will be assessed at baseline, at 3 months and 1 year. The primary outcome is the number of reached cardiovascular health goals (6 metrics) between the interventional group and the group which is treated only by the family physician.

Expected value of the proposed project:

The study has the potential to show that an outpatient rehabilitation program significantly improves vascular risk factors, adherence to medication, enhances quality of life and eventually reduces recurrent strokes and other vascular events. If this is confirmed, introducing outpatient rehabilitation programs will have a major socioeconomic impact.

DETAILED DESCRIPTION:
Background

Stroke represents one of the major health problems worldwide, particularly in transitional and industrialized countries. Stroke ranks first as cause of handicap in adults, second as cause of dementia, third as cause of death and is a frequent cause of epilepsy, depression, falls and acute hospital admissions. Stroke has a remarkable socioeconomic impact, especially in the ageing population, and therefore stroke prevention is important.

Stroke begets stroke. Persons who have suffered a stroke are at high risk of suffering additional strokes. Therefore, prevention in these persons should be part of their medical management. However, secondary stroke prevention is complex due to the numerous risk factors and includes pharmacological interventions and non-pharmacological means for risk factor reduction. Up to 90% of the stroke risk is attributable to vascular risk factors. Therefore, appropriate use of all proven measures of risk factor reduction could prevent up to 90% of all strokes. This includes smoking cessation, control of hypertension and diabetes, anticoagulants or antiplatelet agents and lipid lowering drugs, a healthy lifestyle with regular physical activity, healthy normocaloric diet, moderate or no alcohol consumption, low-normal body weight and avoidance of distress. Importantly, effective stroke prevention can only be achieved by the reduction of several or all vascular risk factors.

Secondary preventive measures and rehabilitation are essential for reduction of recurrent events. Furthermore, moderate to severely handicapped patients should receive in- and outpatient rehabilitation adapted to their individual deficits. The concept of secondary prevention through cardiac rehabilitation is an accepted treatment modality in patients after myocardial infarction or aortocoronary bypass surgery. However, appropriate secondary preventive programs for patients surviving a stroke with minor or no residual deficits are lacking. Therefore, the investigators developed a structured 12 week hospital based out-patient program for stroke patients with minor or no residual deficits based on the already existing format of cardiac rehabilitation to optimize secondary stroke prevention, relieve symptoms, improve neurological functioning, and improve health related quality of life.

In a prospective interventional single center cohort pilot study with 105 patients (that is submitted for publication), the investigators showed that a 12 week outpatient rehabilitation program resulted in a considerable improvement of vascular risk factors, neurological functions, and enhanced health related quality of life (see attached abstract).

The aim of this additional study is to validate the effects of this outpatient program in a prospective, randomized clinical trial with crossover design.

Objective

The aim of this study is to validate the effects of an outpatient secondary prevention program on vascular risk factors, adherence to vascular-protective medication, exercise capacity and health related quality of life.

Methods

This is a prospective, randomized clinical trial. At least 100 patients with minor stroke or transient ischemic attack treated in the University Hospital of Bern will be randomized either to the interventional group or to a group which is treated only by the family physician. All patients will be assessed at baseline, at 3 months and 1 year. The primary outcome is the number of reached cardiovascular health goals (6 metrics: smoking, physical exercise capacity, Mediterranean diet compliance, LDL-Cholesterol, Blood pressure, fasting plasma glucose) between the interventional group and the group which is treated only by the family physician. After inclusion of 100 patients in the study, a study independent statistician will perform a power analysis and the final number of patients to be included will be adapted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic stroke and TIA
* Inclusion in the first 60 days after stroke
* Age between 18 and 75 years
* Minor or no residual neurological deficits (mRS 0-1)
* Written consent by the patient

Exclusion Criteria

* Severe congestive heart failure (NYHA IV)
* Evidence of disabling stroke or dementia as measured by modified Rankin Scale score of ≥3 or a MOCA score < 26
* Any medical condition which disables a patient to participate physical exercise training

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Improvement of a combined endpoint of physical exercise capacity, blood pressure, LDL-cholesterol, HDL-cholesterol, mediterranean diet compliance, and smoking status | 3 months
  The primary endpoint is a combined endpoint of improvement of physical exercise capacity, blood pressure, LDL-cholesterol, HDL-cholesterol, mediterranean diet compliance, and smoking status between the interventional arm and the control arm.

SECONDARY OUTCOMES:
Comparison of neurological function | 3 months
  NIHSS, mRS, 9-Hole-Peg-Test, Functional gait assessment
Comparison of inflammation marker | at 3 months
  C-reactive protein (CRP)
Comparison of adherence to prescribed medication | 3 months
Rate of new diagnosed overseen neurological deficits | 3 months
Comparison of quality-of-life questionnaires | 3 months
  SF 36, DS 14, HADS, Jenkins 4-Items Quest, Fatigue Skala für Motorik und Kognition, EUROQUAL, Stroke Specific Quality of Life, PH Q-9, WHOQQL Bref, Mediterranean Diet Compliance Questionnaire, SWISSPAQ
Comparison of the primary outcome measures between the interventional arm and the control arm | at 3 months, at 12 months
Comparison of drop-out rate between the interventional arm and the control arm | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Simon Jung, MD, Principal Investigator — Department of Neurology, University Hospital of Bern, 3010 Bern, Switzerland
Locations (1):
- Department of Neurology, Bern University Hospital, Bern, Switzerland